CLINICAL TRIAL: NCT00557427
Title: Open-labeled Randomized Comparative Study of the Efficacy and Tolerability of Two Times Daily 250mg Hypericum Versus Once Daily 20 - 40 mg Fluoxetine in Adolescent Patients With Mild to Moderate Depression
Brief Title: Hypericum vs Fluoxetine for Mild to Moderate Adolescent Depression
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Rafa Laboratories (Industry)
Responsible Party: Roy L. Mellovitz, Rafa Laboratories Ltd.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REM-1/MDA; REM-1/MDA
Record Dates: First submitted 2007-11-13; First posted 2007-11-14 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2011-06

CONDITIONS: Depression
Keywords: mild to moderate depression according to the DSM-IV scale
MeSH Terms: conditions — Depression | interventions — Fluoxetine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): hypericum 250mg tablets twice daily for 8 weeks
  Interventions: Drug: hypericum
- B (Active Comparator): fluoxetine 20mg - 40mg daily for 8 weeks
  Interventions: Drug: fluoxetine

INTERVENTIONS:
Drug: hypericum — 250mg tablets twice daily for 8 weeks
  Other Names: Remotiv
  Arms: A
Drug: fluoxetine — 20mg - 40mg daily for 8 weeks
  Arms: B

SUMMARY:
The study is a pilot study where adolescents 12 - 18 years of age with mild to moderate depression will be randomized to receive either hypericum 250mg twice daily or fluoxetine 10mg daily increased to 20mg daily after 1 week and the option to increase to 40mg daily after 4 weeks. Patients will be treated for a total of 8 weeks. Efficacy will be measured using the CDRS-R, BDI-II and the CGI scales. Safety parameters include blood tests, urinalysis and ECG.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Adolescents aged 12 to 18 years
* Patients meeting the criteria for mild to moderate depression according to the DSM-IV scale
* Physical and laboratory examination at baseline compatible with study criteria
* ECG at baseline compatible with study criteria
* Score of at least 40 on the Children's Depression Rating Scale - Revised (CDRS-R) at baseline

Exclusion Criteria:

* Patients with psychosis, bi-polar disease, schizophrenia or significant developmental disorder
* Patients with epilepsy
* Patients with a history of alcohol or substance abuse in the past year
* Initiation of psychotherapy or behavioral therapy in the 2 months prior to screening or during the study.
* Patients who have previously failed to respond to SSRI's or SRNI's
* Patients who have been treated with antidepressants within 2 weeks of screening (4 weeks if fluoxetine)
* Patients with a contraindication to taking either Remotiv or fluoxetine or taking medication contraindicated when taking Remotiv or fluoxetine

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-01; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Rate of clinical response (defined by CDRS-R < 28) at the final/withdrawal visit | 8 weeks

SECONDARY OUTCOMES:
Percentage of patients with a decrease of CDRS-R score > 30 points from baseline | 8 weeks
Final mean CDRS-R score | 8 weeks
Change in CDRS-R score | 8 weeks
Time to clinical response | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Alan Apter, MD, Principal Investigator — Director, child and adolescent division, Schneider Children's Hospital of Israel, Chairman Dept. of Psychiatry Sackler School of Medicine, Tel-Aviv University
Locations (1):
- Schneider Children's Medical Center of Israel, Petah Tikva, Israel

REFERENCES:
- [Result] Findling RL, McNamara NK, O'Riordan MA, Reed MD, Demeter CA, Branicky LA, Blumer JL. An open-label pilot study of St. John's wort in juvenile depression. J Am Acad Child Adolesc Psychiatry. 2003 Aug;42(8):908-14. doi: 10.1097/01.CHI.0000046900.27264.2A. PMID 12874492
- [Result] Simeon J, Nixon MK, Milin R, Jovanovic R, Walker S. Open-label pilot study of St. John's wort in adolescent depression. J Child Adolesc Psychopharmacol. 2005 Apr;15(2):293-301. doi: 10.1089/cap.2005.15.293. PMID 15910213